CLINICAL TRIAL: NCT06064448
Title: A Prospective, Multicenter, Randomized, Parallel and Positive Drug-controlled Clinical Study of Ningbitai Capsule in the Treatment of Chronic Pelvic Pain Syndrome With Erectile Dysfunction
Brief Title: Clinical Observation of Ningmitai Capsule in Treating Chronic Pelvic Pain Syndrome With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xintian Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMT18031S
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Erectile Dysfunction
Keywords: Ningmitai capsule; Sildenafil; Chronic prostatitis/chronic pelvic pain syndrome; Erectile Dysfunction
MeSH Terms: conditions — Prostatitis; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Western Medicine Section (Sildenafil) (Active Comparator): Sildenafil is an effective and commonly used oral PDE5 inhibitor in the treatment of ED.
  In this study, the subjects in the western medicine group will take sildenafil citrate orally, 25mg/capsule, once a night, one capsule each time for 4 weeks.
  Interventions: Drug: Sildenafil
- Traditional Chinese medicine group (Ningmitai capsule) (Experimental): Ningmitai Capsule (Ningmitai®) is Traditional Chinese Medicine which has already used in treatment of Urinary and reproductive system disease (eg. CP/CPPS, ED) in China for more than twenty years.
  In this study, the subjects took Ningmitai Capsule (produced by Guiyang Xintian Pharmaceutical Co., Ltd., Sinopharm Zhunzi Z20025442), 0.38 g/capsule, 3 times a day, 4 capsules each time, and took it after meals for 4 weeks.
  Interventions: Drug: Ningmitai capsule
- Combined group (Ningmitai capsule + sildenafil) (Experimental): In this study, the subjects will take Ningmitai Capsule (produced by Guiyang Xintian Pharmaceutical Co., Ltd., Sinopharm Zhunzi Z20025442), 0.38 g/capsule, 4 capsules each time three times a day, after meals; Sildenafil citrate, 25mg/capsule, once a night, one capsule each time, was taken orally for 4 weeks.
  Interventions: Drug: Ningbitai capsule + sildenafil

INTERVENTIONS:
Drug: Sildenafil — Subjects were given sildenafil citrate, 25mg/capsule, once a night, one capsule each time, for 4 weeks.
  Other Names: Western Medicine Section
  Arms: Western Medicine Section (Sildenafil)
Drug: Ningmitai capsule — The subjects took Ningmitai capsule, 0.38 g/capsule, 3 times a day, 4 capsules each time, after meals, and continued to treat for 4 weeks.
  Other Names: Traditional Chinese medicine group
  Arms: Traditional Chinese medicine group (Ningmitai capsule)
Drug: Ningbitai capsule + sildenafil — The subjects took Ningmitai capsule orally, 0.38 g/capsule, 3 times a day, 4 capsules each time, and took it after meals. Sildenafil citrate, 25mg/capsule, once a night, one capsule each time, was taken orally for 4 weeks.
  Other Names: Combined group
  Arms: Combined group (Ningmitai capsule + sildenafil)

SUMMARY:
Objective: The purpose of this study was to evaluate the clinical efficacy and safety of Ningmitai capsule alone or in combination with sildenafil compared with sildenafil alone in the treatment of CP/CPPS with erectile dysfunction.

Study Design: A multicenter, prospective, randomized and positive drug-controlled clinical study design was adopted.

Interventions:

① Western medicine group (sildenafil): Sildenafil citrate, 25mg/capsule, once a night, one capsule each time, for 4 weeks.

② Chinese medicine group (Ningmitai capsule): Ningmitai capsule, 0.38 g/capsule, 3 times a day, 4 capsules each time, taken after meals for 4 weeks continuously.

③ Combination group (Ningmitai capsule + sildenafil): Ningmitai capsule, 0.38 g/capsule, 3 times a day, 4 capsules each time, taken after meals; Sildenafil citrate, 25mg/capsule, once a night, one capsule each time, was taken continuously for 4 weeks.

DETAILED DESCRIPTION:
Sample size: 214

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 20-50 years;
2. Have a fixed sexual partner and have a normal sexual life;
3. Long-term and repeated pelvic discomfort or pain (NIH-CPSI pain score ≥ 4), or accompanied by lower urinary tract symptoms (micturition score > 4), lasting more than 3 months;
4. Secondary patients with erectile dysfunction after normal erection or sexual intercourse, and IIEF-5 ≤ 21 points;
5. It accords with the main symptoms of damp-heat stagnation syndrome in traditional Chinese medicine;
6. Volunteer subjects and agree to sign informed consent.

Exclusion Criteria:

1. Those who use any antibiotics, α-receptor blockers, PDE5 inhibitors and androgens within one week;
2. Patients with varicocele or tumors in prostate, bladder and urethra;
3. Have received TURP, TUIP, bladder neck incision, transurethral hyperthermia/radiofrequency ablation/balloon dilatation, open prostatectomy, or any other prostate surgery and treatment, such as cryotherapy or hyperthermia;
4. Patients with severe organic ED, drug-induced and traumatic ED, abnormal development of external genitalia or abnormal sex hormone level;
5. Patients with severe cardiovascular and cerebrovascular diseases, liver, kidney and hematopoietic diseases and psychosis;
6. Those who are known to be allergic to the drugs tested in this study or some of their components

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
The response rate of patients at 4 weeks of treatment. | Treatment for 4 weeks
  The response rate is defined as the proportion of patients whose NIH-CPSI pain score decreased by at least 4 points and IIEF-5 score or EHS score increased at 4 weeks of treatment.

SECONDARY OUTCOMES:
NIH-CPSI sub-score and its change value compared with baseline period at 2 weeks and 4 weeks of treatment | Treatment for 2 and 4 weeks
  National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
At 2 and 4 weeks of treatment, IIEF-5 score and its change compared with baseline. | Treatment for 2 and 4 weeks
  Change value = IIEF-5 score after treatment-baseline IIEF-5 score IIEF-5 contains five questions about erectile status, confidence in maintaining erection and satisfaction with sexual intercourse, and is widely used to diagnose ED, judge the severity of ED and evaluate the effectiveness of drug treatment for ED. Total score 25 points, the lower the score, the more serious the symptoms.
The evaluation grade of EHS of patients at 2 weeks and 4 weeks of treatment | Treatment for 2 and 4 weeks
  Erectile hardness score (EHS) is a commonly used method to evaluate the severity of ED in clinic. They are divided into grade I (severe ED), grade II (moderate ED), grade III (mild ED) and grade IV (normal erectile function).

CONTACTS AND LOCATIONS:
Overall Officials: Deng Chunhua, Doctor, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo D, Guo J, Chen T, Liu G, Luo P, Deng Z, Tang YX, Liao Y, Deng C. The efficacy of combination therapy with Ningmitai capsule and sildenafil in men with chronic prostatitis/chronic pelvic pain syndrome and erectile dysfunction: a prospective, multicenter, randomized controlled trial. Sex Med. 2025 May 13;13(2):qfaf024. doi: 10.1093/sexmed/qfaf024. eCollection 2025 Apr. PMID 40365426